CLINICAL TRIAL: NCT06576388
Title: Clinical Trial Evaluating the Safety and Efficacy of EXG001-307 in Patients With Type I Spinal Muscular Atrophy
Brief Title: Clinical Trial to Evaluate the Safety and Efficacy of EXG001-307 in Patients With Spinal Muscular Atrophy Type I
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Hangzhou Jiayin Biotech Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EXG001-307-101
Record Dates: First submitted 2024-08-26; First posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Type I Spinal Muscular Atrophy
MeSH Terms: conditions — Spinal Muscular Atrophies of Childhood

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single Arm-experimental group (Experimental): The dose escalation study included two cohorts with three dose levels: 0.67×1014 vg/kg, 1.1×1014 vg/kg, and 1.5×1014 vg/kg. Among them, the first queue contains two levels, the first dose levels (0.67 x 1014 vg/kg) using the accelerated titration method (i.e. after the first dose levels in group 1 case subjects, when the subjects to 28 days after complete treatment of safety assessment, if not present dose limiting toxicity (DLT), increasing the dose to the next dose levels; Otherwise the study will be terminated .
  Study treatment name:EXG001-307 injection; Dosage form: injection; frequency and duration: single dose
  Interventions: Drug: EXG001-307 injection

INTERVENTIONS:
Drug: EXG001-307 injection — Research process includes filter (subjects signed informed consent for screening period before the pretreatment to the hormone, the longest 28 days), treatment period (the subjects accept including single hormone pretreatment, the study drug infusion) hospitalization and observation and follow-up treatment period (subjects to the participants to 18 months, lost to follow-up, active exit research subjects, or death). Subjects qualified in the screening period entered the treatment period and received EXG001-307, and entered the follow-up period after hospitalization. At the end of the study visit (subject at 18 months of age), eligible subjects will be asked to transfer to the long-term follow-up study.

SUMMARY:
The purpose of this study was to evaluate the safety and preliminary efficacy of a single intravenous injection of exg001-307 in patients with type I spinal muscular atrophy.

The research process includes the screening period (the screening period is from the time the subject signs the informed consent to the time before hormone pretreatment, with a maximum of 28 days), the treatment period (the subject receives hospitalization and observation including hormone pretreatment and single infusion of study drugs), and the follow-up period (the end of the treatment period until the subject reaches the age of 18 months, loss of follow-up, active withdrawal from the study or death). The qualified subjects in the screening period enter the treatment period, receive exg001-307 treatment, and enter the follow-up period after hospitalization observation. At the end of the study visit (subjects 18 months old), eligible subjects will be asked to transfer to the long-term follow-up study.

ELIGIBILITY:
Inclusion Criteria:

1. SMA was diagnosed by bilateral allele SMN1 mutation (deletion or point mutation) gene, and there were 2 copies of SMN2 gene.
2. On the day of administration, the age of the subjects did not exceed the 180th day after birth.
3. The clinical history and signs are consistent with the manifestations of type I SMA, that is, hypotonia, lagging development of motor function, poor head control, round shoulder posture and excessive joint activity.
4. The legal guardian of the subject understands the purpose, possible risks and rights of the test, agrees the subject to participate in the test, completes all research steps, tests and visits, and voluntarily signs the informed consent.
5. During the study period, according to the changes of the subject's condition, the subject's legal guardian was willing to carry out standard treatment requirements such as nasal feeding, noninvasive mechanical ventilation and expectoration machine according to the researcher's suggestions.

Exclusion Criteria:

1. The gestational age at birth was less than 35 weeks (245 days).
2. During the screening period, when the subjects were awake or asleep and did not receive any auxiliary oxygen supply or respiratory support, the blood oxygen saturation was less than 96%.
3. Invasive ventilation or tracheotomy is required, or the current use of noninvasive ventilation support is ≥ 16 hours / day on average.
4. According to the WHO child growth standard (who 2009), the weight is lower than the 3rd percentile by age.
5. Before administration, if the subjects have not been vaccinated or delayed vaccination according to the national vaccination plan of the current month, it will significantly affect their safety according to the evaluation of the researcher and the medical manager of the project team;
6. Active viral infections (including HIV, covid-19, seropositive for hepatitis B or C, torch virus, EBV virus and syphilis).
7. Severe non respiratory diseases within 2 weeks before screening.
8. Upper respiratory tract infection or lower respiratory tract infection within 4 weeks before screening.
9. There are other severe infections or diseases.
10. There are known heart diseases or ECG abnormalities with clinical significance.
11. Known allergy to prednisolone, other glucocorticoids or their excipients.
12. Receive immunosuppressive therapy (e.g. cyclosporin, tacrolimus, methotrexate, cyclophosphamide, intravenous immunoglobulin, rituximab) requiring preventive administration within 3 months before administration.
13. Immunomodulatory drugs (such as thymosin, interferon, etc.) are being used to treat myopathy, neuritis and diabetes (such as immunosuppressive agents, glucocorticoids, insulin).
14. Anti AAV9 antibody titer > 1:50 (determined by ELISA). If the potential subject's anti AAV9 antibody titer > 1:50, it can be retested during the screening period. When the anti AAV9 antibody titer is ≤ 1:50, it can continue to participate in the screening.
15. Abnormal laboratory test values with clinical significance (GGT, ALT and AST > 2.5) × ULN, bilirubin ≥ 3.0 mg / dl, creatinine ≥ 1.0 mg / dl, hemoglobin < 8 or > 18 g / dl; Leukocyte count > 20000 / cm3; Platelet count < 100000 / cm3).
16. Previously participated in clinical research on the treatment of other SMA drugs.
17. Major surgery was expected during study treatment.
18. Other situations that the researcher judges are not suitable to participate in this study.

Max Age: 180 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2022-01-21 (Actual); Primary Completion 2023-09-21 (Actual); Study Completion 2024-01-21 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of EXG001-307 after a single intravenous infusion | up to 18months
  including type and incidence of AE, SAE, AESI, vital signs, physical/neurological examination, immunogenicity, virology, injection/infusion site reactions, 12-lead electrocardiogram, and safety laboratory results recorded

SECONDARY OUTCOMES:
Explore a safe and effective dose range；Assess initial effectiveness； | up to 18 months
  Explore dose limiting toxicity By the time of the study visit at the age of 18 months, the proportion of subjects who could sit alone for ≥ 30 seconds without support was reached according to the Bailey infant development scale version 3 (bsid-iii) Survival at 14 months. Changes in motor function assessment data relative to baseline after 6 months of treatment at the children's Hospital of Philadelphia neuromuscular disease infant test (chop-intend) Proportion of subjects with chop-int score above 40 after 6 months of treatment After 6 months of treatment, the proportion of subjects whose exercise intensity and functional improvement reached development milestones were evaluated according to bsid-iii scale (head control ≥ 3 seconds; sitting alone ≥ 5 seconds without support; sitting alone ≥ 30 seconds without support)

CONTACTS AND LOCATIONS:
Locations (1):
- Hangzhou Jiayin Biotechnology Co., Ltd, Hangzhou, Zhejiang, China